CLINICAL TRIAL: NCT07117513
Title: Heterogeneity Index in Neonatologist-performed Lung Ultrasound in Neonates Receiving Respiratory Support - a Pilot Study
Acronym: NPLUS HI
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Bernhard Schwaberger, Prof. M.D., Medical University of Graz
Other Study IDs: EK1161/2025
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Intensive Care Units, Neonatal; Infant, Newborn; Infant, Premature; Point-of-Care Systems; Ultrasonography; Lung Ultrasound; Lung Ultrasound Score; Image Interpretation, Computer Assisted; Reproducibility of Results; Respiratory Distress Neonatal; Respiratory Support
Keywords: Neonatologist-Performed Lung Ultrasound; Lung Ultrasound; Lung Ultrasound Score; Quantitative Lung Ultrasound; Neonatal Intensive Care Unit; Observer Variability in Imaging; Ultrasound Artifact Interpretation; Respiratory Distress Syndrome in Neonates; respiratory support; preterm neonate; newborn
MeSH Terms: conditions — Premature Birth; Hyaline Membrane Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- term-born neonates and preterm neonates with respiratory support: term-born neonates (37 and more weeks' gestational age) and preterm neonates (28+0-36+6 weeks' gestational age) with respiratory support either invasive or non-invasive admitted to the NICU

SUMMARY:
Lung ultrasound is an increasingly valuable diagnostic tool in neonatal intensive care due to its safety and accessability.

This pilot study investigates whether a quantitative approach - the heterogeneity index, previously only used in fetal lung assessment - can enhance the diagnostic accuracy of neonatologist-performed lung ultrasound (NPLUS). The index will be calculated from raw ultrasound images of preterm and term neonates and compared with conventional lung ultrasound scores to evaluate its clinical relevance.

DETAILED DESCRIPTION:
Lung ultrasound is gaining importance in intensive care medicine, particularly in neonatology, as a rapidly available, and radiation-free alternative to X-ray imaging. Neonatologist-performed lung ultrasound (NPLUS) enables reliable diagnosis of various respiratory conditions in both preterm and term neonates.

It relies on interpreting ultrasound artifacts, pleural line analysis, and detecting consolidations or effusions, thus significantly improving differential diagnosis of neonatal respiratory symptoms. Semi-quantitative lung ultrasound scoring systems have been developed to assess pulmonary aeration patterns and guide clinical decisions-e.g., detecting surfactant deficiency in preterm infants or identifying 'wet lung' in term neonates.

However, subtle sonographic changes related to respiratory symptoms may not be adequately captured on the current 0-3 scale and are subject to interobserver variability. In obstetrics, a heterogeneity index has been introduced to quantitatively assess fetal lung texture with high diagnostic accuracy for postnatal respiratory outcomes.

This study aims to introduce a quantitative ultrasound method into clinical routine to improve diagnostic precision in NPLUS. To our knowledge, this approach has not yet been applied in this context.

In this pilot study, 20 preterm (28+0 to 36+6 weeks) and 20 term (≥37+0 weeks) neonates receiving non-invasive or invasive respiratory support in the NICU will undergo NPLUS at two time points. From the raw ultrasound data, a mean pixel value will be calculated to derive the heterogeneity index, which will then be compared to the traditional lung ultrasound score to assess its clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates born between 28+0 and 36+6 weeks of gestation and term-born neonates (> 37+0 weeks of gestation) admitted to the NICU
* Presence of respiratory distress requiring respiratory support (invasive and non-invasive) at the timepoint of NPLUS 1.
* Written informed consent obtained from the parents prior to the measurement.

Exclusion Criteria:

* cardiopulmonary malformations
* pleural effusion
* pneumothorax

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will include neonates with a gestational age between 28+0 weeks and 42+0 who require either non-invasive or invasive respiratory support in the Department of Neonatology, Medical University Graz, Austria (a tertiary centre).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Determination of the heterogeneity index of NPLUS 1 and NPLUS 2 | one year
  A medical professional will perform the NPLUS (Neontaologist-performed lung ultrasound) at predefined time points after birth: NPLUS 1 within 72 hours of birth and NPLUS 2 within 72 hours (minimum 24 hours) after the first examination.
  The raw ultrasound images will be reviewed by a trained medical professional. A region of interest (ROI) will be manually selected in each lung area that should be analysed. Each ROI will be a square that includes the largest possible area with lung artefacts, starting from the pleura and excluding subcutaneous tissue.
  The grayscale-based analysis will be performed using a custom-made program developed in MATLAB. Texture features in the lung tissue will be related to pathophysiologic processes. The heterogeneity index will then be determined by measuring the intensity of each pixel and calculating the average of all pixel within the ROI.

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Dep. Neonatology, Medical University Graz, Austria, Graz, Styria
  - Medical University Graz, Graz, Styria

IPD SHARING:
Plan to Share IPD: Yes
on request
Supporting Information: Study Protocol
Time Frame: As soon as the recruitment and data analysis are completed, IPD sharing is possible on request (anticipated for May 2026 - August 2026)
Access Criteria: please contact the PI

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT07117513/Prot_SAP_000.pdf